CLINICAL TRIAL: NCT05486715
Title: Vitamin d Level and it's Association With Disease Activity in Egyptian Rheumatoid Arthritis Patients
Acronym: Vitamind
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mariam Samir Farg (Other)
Responsible Party: Sponsor-Investigator, Mariam Samir Farg, Mariam farag, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Vitamin d level
Record Dates: First submitted 2022-03-10; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 65 rheumatoid arthritis patient: Vitamin d effect on rheumatoid arthritis activity on 65 rheumatoid arthritis patients and 65 healthy population
  Interventions: Drug: Vit D
- 65 healthy population: Vitamin d effect on rheumatoid arthritis activity on 65 rheumatoid arthritis patients and 65 healthy population
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — Vit D
  Other Names: Placebo

SUMMARY:
Vitamin D level and its association with disease activity in Egyptian Rheumatoid arthritis (RA) patients

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease that affects about 1% of the human population. Its incidence increases between 25 and 55 years and is the most common type of chronic inflammatory arthritis . It affects joints bilaterally with synovial hyperplasia, cartilage erosion, bone destruction, and progressive loss of function . also characterized by systemic features and joint involvement. It can lead to significant morbidity and mortality so early diagnosis and proper treatment are crucial in decreasing the burden of this disease . According to the World Health Organization mortality database of 31 countries, RA accounts for almost 18% of all deaths caused by different types of arthritis and other musculoskeletal diseases, but the exact cause of RA remains unknown

ELIGIBILITY:
Inclusion Criteria:

* Both males and females in the age group of 1875 years having RA according to the American College of Rheumatology European League Against Rheumatism 2010 criteria (Meena et al., 2018). Will enrolled in this study

Exclusion Criteria:

* Patients with malnutrition, hepatic and renal dysfunction, hyperparathyroidism, hyperthyroidism, diabetes mellitus, and patients on Vitamin D supplementation in the past 6 months or on medications that can affect bone and Vitamin D metabolism (anticonvulsants, diuretics, and thyroxin) were excluded from this study.
* Patients with overlap syndrome
* known allergy to DMARDs, 1,25 dihydroxy vitamin D3 or calcium supplements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Egyptions
Study Population: Sample size was calculated using Epi- Info7. Based on previous study the prevalence of vitamin D insufficiency and deficiency in RA patients was 56% (Cesshetti 2016. ). With a confidence limits of 8% and a confidence level of 80% the minimum number of patients required for this study is 65 patients RA and 65 of healthy
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of vitamin D dificency in Rheumatoid arthritis | 3 years
  prevalence of vitamin D dificency in Rheumatoid arthritis Egyption patients compared by healthy patients

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ab Elmohsen, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No